CLINICAL TRIAL: NCT04284020
Title: Efficacy of Therapeutic Education After Radical Robotic Prostate Surgery: Randomized Clinical Trial
Brief Title: Educational Program Plus Physiotherapy After Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cristina Romojaro Perez, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4/2018
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer; Side Effects
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: two groups: 1 experimental and 1 control group
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational program & pelvic floor muscle training (Experimental): The educational strategy will consist of explaining a healthy lifestyle guide with videos, mobile apps and activities about the anatomy of the pelvic floor and the physiology of the pelvic organs. It will be recommended to avoid risk factors, such as gaining weight, high impact sports, constipation, smoking, or drinking too much caffeine and alcohol. They will also instruct in toilet habits.
  The pelvic floor muscle training (PFMT) protocol will be applied. Participants will perform exercises with anal biofeedback, perineal and erectile dysfunction electrotherapy protocol and surface electromyography. They will perform PFMT in supine position, sitting, standing and walking. The intervention will last 5 weeks, 2 sessions per week. Each session will last 30/40 minutes.
  If the patients have overactive bladder symptoms they will perform transcutaneous tibial nerve stimulation (TTNS) protocol. The intervention will last 5 weeks, 2 sessions per week. Each session will last 30 minutes.
  Interventions: Behavioral: Therapeutic educational program; Other: PFMT; Other: TTNS
- PFMT group (Active Comparator): They will receive a basic behavioral educational strategy in the first session including pelvic anatomy and physiology, recommendations to avoid risk factors and toilet habits.
  The PFMT protocol will be applied. Participants will perform PFMT exercises with anal biofeedback, perineal and erectile dysfunction electrotherapy protocol and surface electromyography. They will perform PFMT in supine position, sitting, standing and walking. The intervention will last 5 weeks, 2 sessions per week. Each session will last 30/40 minutes.
  If the patients have overactive bladder symptoms they will perform transcutaneous tibial nerve stimulation (TTNS) protocol. The intervention will last 5 weeks, 2 sessions per week. Each session will last 30 minutes.
  Interventions: Other: PFMT; Other: TTNS

INTERVENTIONS:
Behavioral: Therapeutic educational program — See arm/group descriptions
  Arms: Educational program & pelvic floor muscle training
Other: PFMT — See arm/group descriptions
  Other Names: Pelvic floor muscle training
Other: TTNS — See arm/group descriptions
  Other Names: Transcutaneous tibial nerve stimulation

SUMMARY:
Objective: to find out the effectiveness of therapeutic education program plus pelvic-perineal physical therapy in radical robotic prostatectomy men in terms of quality of life (QoL), urinary incontinence (UI), erectile dysfunction (ED) and muscle strength.

Design: Randomized, controlled and single blinded clinical trial. Participants will be randomly assigned in two groups. Experimental group: training pelvic-perineal physical therapy plus lifestyle education. Control group: training in pelvic-perineal physical therapy only. In the 2 groups several physical therapy measurements will be undertaken: 1st before physical therapy treatment, 2nd, 3 th and 4th after 3, 6 and 12 months after initial measurement.

Study subjects: Post radical robotic prostatectomy men, which have not been already treated with adjuvant treatment and pelvic-perineal physical therapy, and after reading, understanding and freely signing an informed consent form.

Sample size: 84 subjects will be included (42 subjects per group). To have a statistical power of 90% to detect an average difference of 10 points between two groups in the change of quality of life according to the questionnaire validated in Spanish SF-12, assuming a standard deviation of the change of 20 points based on the study from Hou et al, establishing an alpha risk of 0.05, in a bilateral contrast and assuming a 10% of drops outs.

Data analysis: Separate analyzes of each variable collected in the two groups will be carried out. For continuous variables, means, medians, standard deviations and quartiles will be calculated, depending on the assumption or not, respectively, of the assumption of their normality previously determined with the Shapiro Wilk test (S-W). Qualitative variables will be described with absolute and relative percentage frequencies. Effectiveness will be evaluated by comparing between the two groups of the change in outcome variables between measurements.

ELIGIBILITY:
Inclusion Criteria:

* Men had undergone radical robotic prostate surgery.
* Men reading, understanding and freely signing an informed consent form.

Exclusion Criteria:

* Participants who had received adjuvant therapies (chemotherapy, radiotherapy) before pelvic-perineal physical therapy treatment.
* Men with a history of pelvic organ surgery.
* Men with chronic diseases that affects their quality of life.
* Participants with psychiatric or neurological problems.
* Postoperative men with cognitive limitations to understand information, respond to questionnaires, consent and / or participate in the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in QoL | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  It will be assessed by Short Form 12 (SF-12) Spanish version. The SF-12 consist in 12 items of 8 dimensions: 2 items about physical function, 1 item about social function, 2 items about physical role, 2 items about emotional role, 2 items about mental health, 1 item about vitality, 1 items about body pain, 1 item about general health. The 8 dimensions are scored from 0 (bad health) to 100 (optimal state of health).
Change in UI | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  It will be assessed by International Consultation on Incontinence Questionnaire Urinary Incontinence (ICIQ-UI) Spanish version.
  The ICIQ-UI SF consist in 3 items (Frequency, Quantity and Impact) and 8 questions to identify the UI type. The 3 items are scored from 0 (no incontinence) to 21 (severe incontinence).
  It will be assessed by 1 hour Pad Test. The Pad test consists in weigh a compress after being used under standardized conditions.
Change in Prostatic Symptoms | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  It will be assessed by International Prostate Symptom Score (IPSS) Spanish version.
  The IPSS consist of 6 items plus one about quality of life. The 6 items are scored from 1-7 (mild symptomatology), 8-19 (moderate symptomatology) to 20-35 (severe symptomatology).The item about quality of life is measured qualitatively.
Change in Pelvic Floor Muscle Strength | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  The measuring consists of 4 factors: strength, relax, endurance and repeatability.
  It will be measured with manometry (mmHg).
Change in ED | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  It will be assessed by Short Questionnaire for Erectile Dysfunction (SQUED) Spanish version.
  The SQUED consist of 3 items. The 3 items are scored from 0 (severe dysfunction) to 15 (no dysfunction).
Assess adherence and satisfaction to treatment | 4 measurements to evaluate: before physical therapy treatment, 3 months, 6 months and 12 months after initial measurement.
  It will be assessed by benefit, satisfaction and willingness to continue treatment questionnaire (BSD) Spanish version.
  The BSD consist of 3 items: perception of the benefit, satisfaction with the treatment and willingness of the patient to continue with the treatment.
  The 3 items are scored from 0 (no satisfaction and no adherence) to 10 (much satisfaction and adherence).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Torres-Lacomba, PhD, Study Director — University of Alcalá. FPSM research group. HUPA; Beatriz Navarro-Brázalez, PhD, Study Chair — University of Alcalá. FPSM research group. HUPA
Locations (1):
- University of Alcalá. FPSM research group. HUPA, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No